CLINICAL TRIAL: NCT02581670
Title: Prospective Non-randomized Phase II Study on Stereotactic Body Radiation Therapy for Medically Inoperable Lung and Liver Oligometastases From Breast Cancer
Brief Title: Study on SBRT for Inoperable Lung and Liver Oligometastases From Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, MD, Istituto Clinico Humanitas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1437
Record Dates: First submitted 2015-10-15; First posted 2015-10-21 (Estimated); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer; Metastasis to Liver; Metastasis to Lung
Keywords: oligometastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oligometastatic breast cancer patients (Experimental): Lung and liver stereotactic radiation therapy (SRT) in oligometastatic breast cancer patients medically inoperable, using VMAT RapidArc approach.
  Interventions: Radiation: stereotactic radiation therapy (SRT)

INTERVENTIONS:
Radiation: stereotactic radiation therapy (SRT) — Lung and liver stereotactic radiation therapy (SRT) in oligometastatic breast cancer patients unsuitable for surgery, using VMAT RapidArc approach

SUMMARY:
Investigators designed a phase II study to evaluate safety and efficacy of lung and liver stereotactic radiation therapy (SRT) in oligometastatic breast cancer patients unsuitable for surgery, using VMAT RapidArc approach.

DETAILED DESCRIPTION:
Investigators designed a prospective phase II study to evaluate safety and efficacy of lung and liver stereotactic radiation therapy (SRT) scheduled for oligometastatic breast cancer patients unsuitable for surgery with age major than 18 years old and with adequate performance status (ECOG), using VMAT RapidArc approach. The potential advantage of this technique is the ability to deliver a more selective irradiation to tumour's target while reducing doses to normal tissue, optimizing the therapeutic window.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years with ECOG 0-2
* Diagnosis of Breast Cancer
* DFI (Disease-free interval) > 1 year
* No extrapulmonary and/or extrahepatic disease or other metastatic sites stable or responding after chemotherapy
* No life threatening conditions
* Lung and liver lesions < 5 (with maximum diameter < 5 cm)
* Chemotherapy completed at least 3 weeks before treatment
* Chemotherapy started at least 2 weeks after treatment allowed
* Systemic therapies other than chemotherapy allowed (i.e hormonal therapies and/or immunotherapy)
* Written informed consent

Exclusion Criteria:

* ECOG > 2
* Pregnant women
* Patients with inability to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Toxicity in oligometastatic breast cancer patients monitoring using CTCAE v.4 | 3 years
Local control of disease after SBRT according to EORTC questionnaire | 2 years

SECONDARY OUTCOMES:
Progression free survival using Kaplan-Meyer statistical curves | 2 months
Overall survival using Kaplan-Meyer statistical curves | 2 months
Quality of life at the end of the treatment with questionnaire EORTC QLQ C30 | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Fiorenza De Rose, MD, Principal Investigator — Istituto Clinico Humanitas; Tiziana Comito, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy